CLINICAL TRIAL: NCT03420482
Title: Fecal Microbiota Transplant as Treatment of Hepatic Encephalopathy
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Center for Microbiome Informatics and Therapeutics (Unknown)
Responsible Party: Principal Investigator, Raymond Chung, Principal Investigator, Associate Proffessor of Gastroenterology, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2017P002296
Record Dates: First submitted 2018-01-29; First posted 2018-02-05 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Hepatic Encephalopathy
Keywords: Microbiome; Fecal Microbiota Transplant
MeSH Terms: conditions — Hepatic Encephalopathy | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Intervention Model Description: This is a two part study. The first part is a 10-patient pilot study, used to find 2 stool donors who precipitate the largest improvement in recipient neurological function and microbiome composition. The second part is a 20-patient RCT, where patients will be randomized to FMT or placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomization will be performed by the lab producing the FMT and placebo capsules. Participants, providers, investigators and research assistants will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Fecal Microbiota Transplant (FMT) oral capsules (Experimental): Subjects will receive 15 oral capsules of FMT on days 1, 2, 7, 14, and 21.
  Interventions: Drug: Fecal Microbiota Transplant (FMT) oral capsules
- Placebo capsules (Placebo Comparator): Subjects will receive placebo capsules on the same schedule as the experimental arm (days 1, 2, 7, 14, and 21).
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: Fecal Microbiota Transplant (FMT) oral capsules — Donors will be healthy individuals, selected through a previously published, rigorous screening process. Elizabeth Hohmann M.D. of MGH has demonstrated the safety and therapeutic efficacy of oral frozen FMT capsules in Clostridium difficile infection, and her lab will produce the capsules for this study.
  Arms: Fecal Microbiota Transplant (FMT) oral capsules
Drug: Placebo oral capsule — Oral placebo capsules filled with glycerol and cocoa powder. These capsules are identical in appearance to FMT capsules.
  Arms: Placebo capsules

SUMMARY:
A common complication of advanced liver disease is a condition called hepatic encephalopathy, which leads to confusion. The current treatment options cause side effects, are costly, and do not always work. An abnormal population of bacteria in the intestines may be causing this condition, and transplanting bacteria from the colon of a healthy person may treat it. In this research study, the investigators will first find two healthy stool donors whose stool donation improves the gut bacteria of patients with advanced liver disease and helps them think more clearly. Then, in a randomized controlled trial, the investigators will compare the ability of stool donation from these two best donors versus a placebo to improve the neurological function of patients with advanced liver disease. If the investigators find the expected results, there will be a new effective therapy for patients with advanced liver disease and the very troublesome complication of hepatic encephalopathy.

DETAILED DESCRIPTION:
Decades of investigation demonstrate that hepatic encephalopathy (HE), a common complication of cirrhosis characterized by impaired cognition, develops as a consequence of intestinal microbial products reaching the brain. Recent investigation has found that cirrhotic patients, especially those who have developed HE, have intestinal dysbiosis compared to normal controls. Several plausible mechanisms explain how intestinal dysbiosis could lead to HE. There is limited prior literature on the efficacy of FMT in cirrhosis. The largest documented study of 10 cirrhotic patients receiving a single FMT enema found no significant change in microbiome diversity as assessed by 16S rRNA sequencing. The investigators hypothesize that aggressive manipulation of the microbial composition with fecal microbiota transplant (FMT) will improve neurological function in patients with a history of cirrhosis and HE. The investigators additionally hypothesize that five oral FMT capsule administrations from a previously efficacious stool donor will significantly change the intestinal microbiome composition of a cirrhotic patient. The study will consist of a 10-patient open-label pilot study to identify efficacious stool donors, defined as donors who precipitate the largest improvement in recipient neurological function and microbiome composition. The two most efficacious pilot study stool donors will be selected to donate stool for the randomized controlled trial (RCT). The 20-patient RCT will investigate the effect of FMT on neurological outcomes in patients with cirrhosis and a history of HE. Subjects will be randomized to receive 5 doses of oral FMT capsules or placebo capsules over 21 days. Cognitive testing and stool collections will occur at 4 time points, to assess for changes in neurological function and microbiome composition. The primary outcome is change in neurological function after FMT. The main secondary outcome is change in microbiome composition after FMT. This study could provide valuable information about the ability of FMT to improve intestinal dysbiosis in cirrhosis and treat HE.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cirrhosis: Based on liver biopsy or clinical assessment of a hepatologist based on history, exam, laboratory and radiographic evidence
* History of at least one episode of overt HE, defined by West Haven Criteria Grades II to IV; episodes of HE that were precipitated by gastrointestinal hemorrhage requiring transfusion of at least 2 units of blood, by medication use, by renal failure requiring dialysis, or by injury to the central nervous system will not be counted as previous HE episodes
* Compliant with lactulose and rifaximin treatment (lactulose: at least one dose at least 5 days per week; rifaximin: at least one dose at least 5 days per week)

Exclusion Criteria:

* Current episode of overt HE as defined by West Haven Criteria Grades II to IV
* Expectation of liver transplantation within two months of the screening visit
* Current infection
* Variceal bleeding in the last 4 weeks
* Gut-absorbable or intravenous antibiotic therapy (including ciprofloxacin for SBP prophylaxis) in the last 3 months
* Alcohol or illicit drug intake within 3 months, by history and available serum testing; alcohol use will be characterized as >1 alcoholic drink / month
* PSC as etiology of liver disease, as prior literature has suggested these individuals have a unique microbiome
* History of Roux-en-Y Gastric bypass
* On immunosuppressive medications
* Positive C. difficile test
* Scoring above a threshold cut-off on the Psychometric Hepatic Encephalopathy Score (PHES)
* MELD > 17
* History of spontaneous bacterial peritonitis
* History of low ascites protein ( ≤ 1g/dL) in the last year
* Hemodialysis in the last 30 days
* Other significant laboratory abnormalities: serum creatinine > 2.0 mg/dL, hemoglobin < 8 g/dL, serum sodium < 125 mmol/L, serum calcium > 11.0 mg/dL, serum potassium < 2.5 mmol/L
* Placement of a portosystemic shunt or transjugular intrahepatic portosystemic shunt
* Unstable doses of opiates, benzodiazepines or other sedating medication
* Unable to provide consent; a. If MMSE is < 18 or the patient is deemed to not have capacity by an investigator, a legally authorized representative (surrogate) will be allowed to provide consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-04-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Psychometric Hepatic Encephalopathy Score (PHES) | Before the first administration of FMT (day 0) and one week after the last administration of FMT (day 28)
  The PHES is a validated assessment tool specifically designed for HE trials to test cognitive and psychomotor processing speed and visuomotor coordination. The PHES is a battery of 5 pencil-paper tests, completed in 15-20 minutes. The primary outcome is the change in PHES score from immediately before FMT to 1 week after the last dose of FMT.

SECONDARY OUTCOMES:
Adverse events | Adverse event reporting will take place on day 2, 4, 7, 14, 21, then 1, 4 weeks after the last FMT administration.
  Adverse events will be graded based on CTCAE V.4.03.
Stroop Test | Before the first administration of FMT (day 0) and one week after the last administration of FMT (day 28)
  The Stroop Test evaluates psychomotor speed and cognitive flexibility by the interference between recognition reaction time to a colored field and a written color name. A smartphone application software called "EncephalApp Stroop Test" will be used, validated to identify cognitive dysfunction in cirrhosis and screen for covert hepatic encephalopathy.
36-Item Short Form Health Survey (SF-36) | Before the first administration of FMT (day 0) and one week after the last administration of FMT (day 28)
  The SF-36 is a highly utilized quality of life questionnaire. There are 8 health concepts assessed by the survey, which includes physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions. Each of these health concepts is scored on a scale from 0 to 100. 0 is considered the worst outcome and 100 is considered the most favorable health state on each subscale. There will be no total or summed score.
Ammonia level | Before the first administration of FMT (day 0) and one week after the last administration of FMT (day 28)
  Ammonia is a serology with a known association with hepatic encephalopathy.
Microbiome engraftment | Before the first administration of FMT (day 0), after 3 FMT administrations (day 14), one week after the last administration of FMT (day 28) and 4 weeks after the last administration of FMT.
  Sequence-based microbiome surveys will be carried out using metagenomic sequencing. Computational analyses will investigate donor microbiota colonization by comparing single-nucleotide variants in strain level data between the donor and recipient.

CONTACTS AND LOCATIONS:
Overall Officials: Raymond T Chung, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Bajaj JS, Kassam Z, Fagan A, Gavis EA, Liu E, Cox IJ, Kheradman R, Heuman D, Wang J, Gurry T, Williams R, Sikaroodi M, Fuchs M, Alm E, John B, Thacker LR, Riva A, Smith M, Taylor-Robinson SD, Gillevet PM. Fecal microbiota transplant from a rational stool donor improves hepatic encephalopathy: A randomized clinical trial. Hepatology. 2017 Dec;66(6):1727-1738. doi: 10.1002/hep.29306. Epub 2017 Oct 30. PMID 28586116
- [Background] Youngster I, Mahabamunuge J, Systrom HK, Sauk J, Khalili H, Levin J, Kaplan JL, Hohmann EL. Oral, frozen fecal microbiota transplant (FMT) capsules for recurrent Clostridium difficile infection. BMC Med. 2016 Sep 9;14(1):134. doi: 10.1186/s12916-016-0680-9. PMID 27609178
- [Background] Kao D, Roach B, Silva M, Beck P, Rioux K, Kaplan GG, Chang HJ, Coward S, Goodman KJ, Xu H, Madsen K, Mason A, Wong GK, Jovel J, Patterson J, Louie T. Effect of Oral Capsule- vs Colonoscopy-Delivered Fecal Microbiota Transplantation on Recurrent Clostridium difficile Infection: A Randomized Clinical Trial. JAMA. 2017 Nov 28;318(20):1985-1993. doi: 10.1001/jama.2017.17077. PMID 29183074
- [Derived] Bloom PP, Donlan J, Torres Soto M, Daidone M, Hohmann E, Chung RT. Fecal microbiota transplant improves cognition in hepatic encephalopathy and its effect varies by donor and recipient. Hepatol Commun. 2022 Aug;6(8):2079-2089. doi: 10.1002/hep4.1950. Epub 2022 Apr 5. PMID 35384391